CLINICAL TRIAL: NCT03401502
Title: A TSHRN1201 Sub-study-To Evaluate the Effects of add-on Ranolazine on Exercise Tolerance and Angina Frequency in Patients With Stable Angina Pectoris.
Brief Title: A TSHRN1201 Sub-study-To Evaluate the Effects of add-on Ranolazine on Exercise Tolerance and Angina Frequency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TSH Biopharm Corporation Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSHRN1701
Record Dates: First submitted 2018-01-07; First posted 2018-01-17 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Angina
MeSH Terms: conditions — Angina Pectoris | interventions — Ranolazine

STUDY DESIGN:
Intervention Model Description: * Treatment group:Ranolazine 1000 mg:
  * Control group: Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment groups (Experimental): Ranolazine 1000 mg
  Interventions: Drug: Ranolazine
- Control group (Placebo Comparator): Placebos
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Ranolazine — Oral, b.i.d
  Other Names: RNTA
  Arms: Treatment groups
Drug: Placebos — Oral, b.i.d
  Other Names: Placebo
  Arms: Control group

SUMMARY:
This is a double-blind, randomized, placebo-controlled, and parallel study. The study is comprised of three main phases: a single-blind placebo run-in qualifying phase lasting about 14 days, a double-blind treatment phase of 12 weeks, and a 2-week follow-up phase. Approximately 18 patients will be enrolled and randomly assigned to receive placebo or 1,000 mg of extended-release Ranolazine twice-daily for 12 weeks to reach 14 evaluable patients at the end of the study.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled, and parallel study. The study is comprised of three main phases: a single-blind placebo run-in qualifying phase lasting about 14 days, a double-blind treatment phase of 12 weeks, and a 2-week follow-up phase. Approximately 18 patients will be enrolled and randomly assigned to receive placebo or 1,000 mg of extended-release Ranolazine twice-daily for 12 weeks to reach 14 evaluable patients at the end of the study.

Patients with chronic angina pectoris will be screened for eligibility after providing informed consent. Patients present with the symptoms of stable angina after withdrawn from other antianginal agents and given the required background therapy for at least 5 days will be qualified for entering this study and performing 1st ETT qualifying test.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥ 20 years old.
2. A minimum 3-month history of stable angina.
3. Patients with diagnosis of coronary artery disease (CAD) via at least one of the following criteria:

   * Angiographic evidence of ≥ 50% stenosis of ≥ 1 major coronary artery;
   * CT angiographic evidence of ≥ 50% stenosis of ≥ 1 major coronary artery;
   * History of previous myocardial infarction (MI)*;

     *Previous MI history of patients has to be occurred and diagnosed at least 2 months prior entering this study.
   * A stress-induced reversible perfusion defect identified by radionuclide or echocardiographic imaging.
4. Patients present with the symptoms of stable angina after withdrawn from other antianginal drugs and given the required background therapy for at least 5 days will be qualified for entering this study and performing 1st ETT qualifying test.
5. Patients developed exercise-induced ECG ischemia during two qualifying exercise treadmill tests. The difference between twotests should be ≤ 20% of the longer test or ≤ 1 minute.
6. Willing and able to provide a written informed consent.

Exclusion Criteria:

1. Factors that might compromise ECG or ETT interpretation.

   * Patients with resting ST-segment depression ≥ 1mm in any lead.
   * Left bundle-branch block.
   * Patients implanted with pacemaker.
   * Patients under Digitalis therapy.
2. Patients with family history of (or congenital) long QT syndrome.
3. Patients with congenital heart disease.
4. Patients with uncorrected valvular heart disease.
5. Patients with unstable angina, or MI, or coronary revascularization procedure ≤ 2 months prior enter this study.
6. Female who is pregnant/lactating or planning to be pregnant, or female of childbearing potential* who is not using medically recognized method of contraception.

   *Other than those who have been surgically sterilized (defined as having undergone hysterectomy or bilateral oophorectomy or bilateral salpingectomy; tubal ligation alone is not considered sufficient) or one year post-menopausal.
7. Patients are under any one of the following conditions:

   * New York Heart Association (NYHA) Class III or Class IV congestive heart failure (CHF);
   * QTc > 450 msec at screening;
   * Active myocarditis, pericarditis, hypertrophic cardiomyopathy;
   * Uncontrolled hypertension (defined as SBP > 180 mmHg). Voltage criteria for left ventricular hypertrophy in the absence of repolarization abnormalities will not be exclusion criteria.
8. Use of any investigational product ≤ 4 weeks prior to screening.
9. Patients with severe hepatic disease (e.g., liver cirrhosis).
10. Patients with impaired renal function (defined as serum Cr >1.5 mg/dl).
11. Patients with any condition or disease which is considered not suitable for this study by investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
ETT performing duration | at trough (12 hours after dosing) at Week 12
  To compare the change from baseline of ETT performing duration between add-on Ranolazine and placebo

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng Dist, Taiwan

IPD SHARING:
Plan to Share IPD: No